CLINICAL TRIAL: NCT06552728
Title: The Effects of Energy Healing in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Richard Edmund Harris, Samueli Endowed Chair and Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5179
Record Dates: First submitted 2024-08-06; First posted 2024-08-14 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibromyalgia participants - Energy Healing Intervention (Experimental): Female Fibromyalgia patients ages 18-75 who meet inclusion/exclusion criteria as stated in the IRB approved study protocol.
  Interventions: Other: Energy Healing

INTERVENTIONS:
Other: Energy Healing — EH derives from the theory that by using the body's biological energy, there can be a therapeutic effect that guides the patient towards a homeostatic state. Preliminary data in chronic pain patients, suggests that EH, delivered by an experienced practitioner, is able to reduce self-reported pain symptoms within minutes. Effects lasting for weeks to months have also been anecdotally reported. For patients with pain, this can result in a reduction of symptoms. Participants will also be presented with sham EH as a control.

SUMMARY:
This study aims to study the clinical effects of Energy Healing using fMRI and determine its application to Fibromyalgia patients. We also want to find out how active Energy Healing compares to sham Energy Healing in terms of brain connectivity and pain interference scores.

DETAILED DESCRIPTION:
The primary objective is to investigate the effects of energy healing as compared to sham EH on brain connectivity of the insula/salience network, sensory motor network, and default mode network as primary outcomes using fcMRI.

The secondary objective is to evaluate the effectiveness of EH in reducing clinical pain severity and interference (secondary outcomes) and their relationship to brain connectivity (secondary outcomes) as compared to placebo/sham EH.

The exploratory objective is to understand the effects of EH versus sham EH on brain functional response to visual stimuli, insular glutamate, heart rate variability, mood, sleep, and fatigue symptoms in fibromyalgia patients (all exploratory outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 and under 75 years of age.
* Fibromyalgia patients must meet the 2016 Fibromyalgia Diagnostic Criteria for the classification of FM.
* Mean recalled pain over the last seven days (7-day recall) between 4-10 cm on Visual - - - - Analog Scale (VAS) for pain with no pain free days in the last 2 months and active pain in resting state lying on back.
* No contraindications for MRI, such as metal in the body or electrical devices in the body.
* Willing to limit the introduction of any new medications or treatment modalities for control of FM symptoms during the study.
* Able to travel to the study site to receive MRI, EH, and sham EH sessions up to twice weekly.
* Understanding and willing to complete all study procedures.
* Capable of giving written informed consent.
* Proficient ability to speak, read, and write in english.

Exclusion Criteria:

* EH within the last 6-months.
* Have received past treatment from Charlie Goldsmith or know of him or his work.
* Contraindications to MRI and fcMRI methods. These may include but are not limited to: surgical clips, surgical staples, metal implants, and certain metallic dental material, claustrophobia, etc. [Note: a more formal description of contraindications for MRI is present -in our DSM Plan].
* Presence of known past procedures, devices in the body, claustrophobia, or other contraindications for MRI
* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain.
* Peripheral neuropathy that interferes with activities of daily living.
* Routine daily use of narcotic analgesics or history of substance abuse.
* Stimulant medications, such as those used to treat ADD/ADHD (e.g., amphetamine/ dextroamphetamine [Adderall®], methylphenidate, dextroamphetamine), or the fatigue associated with sleep apnea or shift work (e.g., modafinil), are excluded.
* Concurrent participation in other therapeutic trials.
* Pregnant or nursing.
* Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation).
* Active substance abuse disorder in the past 24 months as determined by subject self-report.
* Use of PRN over the counter (OTC) pain medications (NSAIDs, etc.) on day of MRI scan.
* Use of PRN narcotic pain medication 48 hours prior to MRI scan.
* Current active litigation for FM pain.
* Any impairment, activity or situation that in the judgment of the Principal Investigator or other team member that would prevent satisfactory completion of the study protocol. This includes unreliable, or inconsistent pain scores as deemed by the principal investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Neural connectivity | Pre screening, Baseline, Intervention, 3- and 6-month follow ups Post-treatment
  change in brain connectivity of the insula/salience network (SLN), sensory motor network (SMN), and default mode network (DMN) resulting from energy healing (EH) as compared to sham EH.

SECONDARY OUTCOMES:
Pain severity | Pre screening, Baseline, Intervention, 3- and 6-month follow ups Post-treatment
  changes in pain severity and interference and their relationships to brain connectivity. We will determine if EH is effective in reducing clinical pain severity and interference as compared to placebo/sham EH and assess changes in their relationships before and after EH/sham EH to changes in brain connectivity.
Effects of Energy Healing vs sham Energy Healing on brain functional response | Pre screening, Baseline, Intervention, 3- and 6-month follow ups Post-treatment
  As exploratory outcomes, we will also explore the effects of EH vs sham EH on brain functional response to visual stimuli, insular Glx, heart rate variability, mood, sleep, and fatigue symptoms in FM patients.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Harris, PhD, Principal Investigator — UCI SSIHI
Locations (1):
- University of California at Irvine, Irvine, California, United States